CLINICAL TRIAL: NCT01715194
Title: Telemedicine to Enhance Adherence to Continuous Positive Airway Pressure Therapy in Patients With Obstructive Sleep Apnea Syndrome; a Randomized Placebo-controlled Prospective Study
Brief Title: Telemedicine to Enhance Adherence to CPAP Therapy in Patients With OSAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Otto D. Schoch (Other)
Responsible Party: Sponsor-Investigator, Otto D. Schoch, Sponsor investigator, Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EKSG 12/076
Record Dates: First submitted 2012-10-10; First posted 2012-10-26 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: OSAS; CPAP; Adherence; Telemedicine
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telemedicine intervention (Active Comparator): In the telemedicine intervention arm, a telemetry device is instructed and attached to the CPAP. Patients are instructed to use CPAP every night. Data of the CPAP are downloaded to the internet once daily. On week days, a nurse is checking the downloaded data three times per week. The nurse contacts the patient if
  1. CPAP was used <4h/ night for 2 consecutive night
  2. the median leakage was above 0.4 L/sec on 2 consecutive nights The nurse informs the patient of the problem observed, asks for explanations and gives advice on possibilities to solve the problem. The common problems and the respective solutions are discussed according to the ELF facts sheet (Dry mouth/throat, nasal congestion, skin irritation, conjunctivitis, headache, loss of benefits, appendix 1). The patient is encouraged to use CPAP every night. In the case of regular use and acceptable leakage, a congratulatory message is sent to the patient via sms or e-mail (for procedural rules, see appendix 4).
  Interventions: Device: Telemedicine intervention
- Control (without telemedicine) (No Intervention): In the control arm, no device is attached to the CPAP machine, but data stored in the CPAP machine are collected at the follow-up visit after 1 month of CPAP use.

INTERVENTIONS:
Device: Telemedicine intervention — Patients undergoing telemedicine intervention
  Other Names: ResMed Telemedicine S9 Wireless-Modul
  Arms: Telemedicine intervention

SUMMARY:
We hypothesize that the use of telemedicine combined with support interventions by short messages, telephone calls and ambulatory visits to control CPAP treatment during the first month improves adherence and reduces unresolved side effects of therapy.

The primary objective of an OSAS treatment program is to successfully implement indicated CPAP in the highest possible proportion of patients in order to lower the proportion of untreated OSAS in the population. On an individual basis, it has been shown that a longer duration of CPAP use is associated with better outcomes in terms of daytime functioning and in the control of metabolic and blood pressure effects of CPAP. For our study, we have therefore decided to use 2 co-primary endpoints, taking into account both aspects of adherence mentioned. Cardiovascular complications are a major concern in OSAS patients. Effective CPAP treatment has been shown to reduce surrogate measures of cardiovascular risk. We hypothesize that intensified efforts for CPAP adherence with telemedicine has a positive impact on a number of surrogate measures of the cardiovascular risk at 1 and 6 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic OSAS patients with an AHI and an oxygen desaturation index (ODI) of >5/h in polysomnography (PSG) consenting to start longterm CPAP treatment.

Exclusion Criteria:

* Age <18 years
* Unable to communicate in German, English, French or Italian
* Alcohol consumption > 4 units >4 times a week
* Acute manifestation of psychiatric diseases
* Life expectancy of < 6 months for any reason
* Surgical obesity treatment planned within the next 6 months
* Predominantly Central sleep apnea and cheyne stokes respiration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2012-12; Primary Completion 2015-12 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Proportion of nights with CPAP use (defined as ≥1h of CPAP use per night within the last month including nights of no-use of CPAP) at 6 months | at 6 months

SECONDARY OUTCOMES:
Average nightly use of CPAP during the first 6 months of treatment (minutes per night including nights of no-use of CPAP since day 1) | at 6 months

OTHER OUTCOMES:
Proportion of nights with efficient CPAP use (defined as ≥4h of CPAP use per night within the last month including nights of no-use of CPAP) at 6 months | at 6 months
Average nightly use of CPAP during the first 6 months of treatment (minutes per night excluding nights of no-use of CPAP) | at 6 months
Proportion of CPAP users (defined as ≥1h of CPAP use per night within the last week) at 1 month | at 1 month
Average nightly use of CPAP during the first month of treatment (minutes per night including nights of no-use of CPAP since day 1) | at 1 month
Proportion of efficient CPAP users (defined as ≥4h of CPAP use per night within the last week including nights of no-use of CPAP) at 1 month | at 1 month
Average nightly use of CPAP during the first month of treatment (minutes per night excluding nights of no-use of CPAP) | at 1 month
Mask leakage at 1 and 6 months | at 1 and 6 months
Adverse effects on CPAP at 1 and 6 months | at 1 and 6 months
  The proportion of patients with insomnia/dyssomnia due to CPAP, skin problems due to the mask, oronasal dryness or other treatment related complaints is assessed.
Patient satisfaction (measured with a specifically designed short questionnaire and on a visual analogue scale (VAS)) at 1 and 6 months | at 1 and 6 months
Likelihood of discontinuing CPAP is estimated with Kaplan Meyer analysis and groups are compared with the Cox proportional hazard ratio analysis. | at 6 months
Cardiovascular risk factors in serum (e.g. cholesterol, C-peptid, ...), blood pressure and night time assessment of sleep quality with the novel assessment tool "SOMNOcheck micro". | at 1 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Martin Brutsche, MD, PhD, Study Director — Cantonal Hospital of St. Gallen
Locations (1):
- Cantonal Hospital St. Gallen, Sankt Gallen, CH, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sparrow D, Aloia M, Demolles DA, Gottlieb DJ. A telemedicine intervention to improve adherence to continuous positive airway pressure: a randomised controlled trial. Thorax. 2010 Dec;65(12):1061-6. doi: 10.1136/thx.2009.133215. Epub 2010 Sep 29. PMID 20880872
- [Background] Lankford DA. Wireless CPAP patient monitoring: accuracy study. Telemed J E Health. 2004 Summer;10(2):162-9. doi: 10.1089/tmj.2004.10.162. PMID 15319046
- [Background] Smith CE, Dauz ER, Clements F, Puno FN, Cook D, Doolittle G, Leeds W. Telehealth services to improve nonadherence: A placebo-controlled study. Telemed J E Health. 2006 Jun;12(3):289-96. doi: 10.1089/tmj.2006.12.289. PMID 16796496
- [Background] Stepnowsky CJ, Palau JJ, Marler MR, Gifford AL. Pilot randomized trial of the effect of wireless telemonitoring on compliance and treatment efficacy in obstructive sleep apnea. J Med Internet Res. 2007 May 17;9(2):e14. doi: 10.2196/jmir.9.2.e14. PMID 17513285
- [Background] Kwiatkowska M, Ayas N. Can telemedicine improve CPAP adherence? Thorax. 2010 Dec;65(12):1035-6. doi: 10.1136/thx.2010.140897. Epub 2010 Oct 26. No abstract available. PMID 20978030
- [Derived] Schoch OD, Baty F, Boesch M, Benz G, Niedermann J, Brutsche MH. Telemedicine for Continuous Positive Airway Pressure in Sleep Apnea. A Randomized, Controlled Study. Ann Am Thorac Soc. 2019 Dec;16(12):1550-1557. doi: 10.1513/AnnalsATS.201901-013OC. PMID 31310575